CLINICAL TRIAL: NCT01316653
Title: Growing Right Onto Wellness (GROW): Changing Early Childhood Body Mass Index (BMI) Trajectories
Acronym: GROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Nashville Metro Parks and Recreation Department (Unknown); Nashville Public Library Foundation (Unknown)
Responsible Party: Principal Investigator, Shari Barkin, MD, MSHS, William K. Warren Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100591; 5U01HL103620-03 (NIH)
Record Dates: First submitted 2011-03-03; First posted 2011-03-16 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Overweight and Obesity; Childhood Obesity
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROW Smarter (Active Comparator): Library based program to promote early literacy
  Interventions: Behavioral: GROW Smarter
- GROW Healthier (Experimental): Healthy lifestyle intervention focused on building healthy lifestyle skills for preschool children and participating parents and building new social networks between the intervention group members.
  Interventions: Behavioral: GROW Healthier; Behavioral: GROW Smarter

INTERVENTIONS:
Behavioral: GROW Healthier — Group sessions that meet once weekly for 3 months (intensive phase) with choice of phone call session as preferred by participant, phone call coaching monthly for 9 months (maintenance phase), and monthly cues to action to use one's built environment for healthy activities for 24 months (sustainability phase)
  Arms: GROW Healthier
Behavioral: GROW Smarter — Group sessions that meet six times over the course of three years with quarterly newsletters.

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial that examines how a family based, community centered intervention effects early childhood BMI trajectories.

DETAILED DESCRIPTION:
Increases in sedentary lifestyle and high calorie food consumption, among other factors, have contributed to epidemic levels of childhood obesity in the US. Children who are overweight during the preschool period are more likely to become overweight adolescents and obese adults. Food preferences and activity habits set in early childhood can profoundly influence lifelong trajectories for Body Mass Index (BMI) and health. Specifically, rapid BMI gain in early childhood has been established to affect adulthood mortality and morbidity. Unfortunately, the longer such unhealthy patterns are in place, the more difficult it can be to reverse them. Therefore, healthy lifestyle interventions targeted at children as early as preschool have enormous potential to affect lifelong health. Furthermore, nutrition and activity patterns are determined not only at the child level, but within the family and the community.

This study will assess the impact of a family-based and community centered multilevel behavioral intervention addressing nutrition and physical activity with high risk parent-preschool children dyads to promote pediatric obesity prevention. The 7 year study will follow 600 parent preschool child dyads, half of whom will be randomized into the intervention condition which will utilize a health literate approach, build new social networks, utilize behavior modification tools including goal setting, self monitoring, and problem solving, and create behavior-environmental synergy with cues to action for use of the built environment for healthy behaviors. Both the intervention and control group (separately) will receive the control condition in which parent-child dyads will receive a literacy promotion/school success curriculum.

The primary outcome of interest will be early childhood BMI trajectories measured at multiple time points over the three year RCT. Additional measures collected throughout the study from children and parents will include: tricep skin fold, waist circumference, actigraphy, 3-day diet recalls, questionnaires, social network data, and saliva to assess a genetics/epigenetics associated with obesity. Consistent with a multilevel systems approach, the investigators will develop and assess built environment changes related to obesity prevention. Moreover, working with the study's community partners, the investigators will evaluate how this approach affects local policy.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Address in select zip code regions around participating Metro community centers
* Parental commitment to consistent participation
* Consistent phone access for 3 years
* Child aged 3-5 years old
* Child BMI ≥ 50% and < 95% (no diagnosis of failure to thrive or difficulty with appropriate weight gain)
* Healthy parent and child (without medical conditions necessitating limited physical activity)
* Parent ≥ 18 years of age

Exclusion Criteria:

* Non English or Spanish speaking
* Address outside select zip code regions around participating Metro community centers
* Lack of parental commitment to consistent participation
* Lack of consistent phone access
* Child outside specified age range
* Child BMI < 50% or ≥ 95%
* Parents and/or children who are diagnosed with medical illnesses where regular exercise might be contraindicated
* Parent < 18 years of age

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 610 (Actual)
Dates: Start 2011-06; Primary Completion 2017-06-13 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Early Childhood BMI Trajectory | Baseline, 3 months, 9 months, 12 months, 24 months, and 36 months

SECONDARY OUTCOMES:
Average daily energy intake (kcal) | Baseline, 12 months, 24 months, and 36 months
Percentage of Energy Intake from Fat | Baseline, 12 months, 24 months, and 36 months
Percentage of Energy Intake from Carbohydrates | Baseline, 12 months, 24 months, and 36 months
Percentage of Energy Intake from Protein | Baseline, 12 months, 24 months, and 36 months
Average daily time (minutes) spent in rest and sedentary behavior | Baseline, 12 months, 24 months, and 36 months
Average daily time (minutes) spent in moderate and vigorous physical activity | Baseline, 12 months, 24 months, and 36 months
Parent community center use with child | Baseline, 12 months, 24 months, and 36 months
  never versus at least once
Parent BMI | Baseline, 3 months, 9 months, 12 months, 24 months, and 36 months
Parent Waist Circumference | Baseline, 12 months, 24 months, and 36 months
Parent Triceps Skinfold | Baseline, 12 months, 24 months, and 36 months
Child Waist Circumference | Baseline, 12 months, 24 months, and 36 months
Child Triceps Skinfold | Baseline, 12 months, 24 months, and 36 months

OTHER OUTCOMES:
Social Network | Baseline, 3 months, 12 months, and 36 months
  Ties between participants

CONTACTS AND LOCATIONS:
Overall Officials: Shari Barkin, MD, MSHS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Heerman WJ, Bian A, Shintani A, Barkin SL. Interaction between maternal prepregnancy body mass index and gestational weight gain shapes infant growth. Acad Pediatr. 2014 Sep-Oct;14(5):463-70. doi: 10.1016/j.acap.2014.05.005. PMID 25169157
- [Background] Ruiz RM, Tracy D, Sommer EC, Barkin SL. A novel approach to characterize physical activity patterns in preschool-aged children. Obesity (Silver Spring). 2013 Nov;21(11):2197-203. doi: 10.1002/oby.20560. Epub 2013 Oct 17. PMID 24136917
- [Background] Gesell SB, Barkin SL, Valente TW. Social network diagnostics: a tool for monitoring group interventions. Implement Sci. 2013 Oct 1;8:116. doi: 10.1186/1748-5908-8-116. PMID 24083343
- [Background] Po'e EK, Heerman WJ, Mistry RS, Barkin SL. Growing Right Onto Wellness (GROW): a family-centered, community-based obesity prevention randomized controlled trial for preschool child-parent pairs. Contemp Clin Trials. 2013 Nov;36(2):436-49. doi: 10.1016/j.cct.2013.08.013. Epub 2013 Sep 5. PMID 24012890
- [Background] Reinert KR, Po'e EK, Barkin SL. The relationship between executive function and obesity in children and adolescents: a systematic literature review. J Obes. 2013;2013:820956. doi: 10.1155/2013/820956. Epub 2013 Feb 21. PMID 23533726
- [Background] White RO, Thompson JR, Rothman RL, McDougald Scott AM, Heerman WJ, Sommer EC, Barkin SL. A health literate approach to the prevention of childhood overweight and obesity. Patient Educ Couns. 2013 Dec;93(3):612-8. doi: 10.1016/j.pec.2013.08.010. Epub 2013 Aug 19. PMID 24001660
- [Background] Gesell SB, Barkin SL, Sommer EC, Thompson JR, Valente TW. Increases in Network Ties Are Associated With Increased Cohesion Among Intervention Participants. Health Educ Behav. 2016 Apr;43(2):208-16. doi: 10.1177/1090198115599397. Epub 2015 Aug 17. PMID 26286298
- [Background] Heerman WJ, Krishnaswami S, Barkin SL, McPheeters M. Adverse family experiences during childhood and adolescent obesity. Obesity (Silver Spring). 2016 Mar;24(3):696-702. doi: 10.1002/oby.21413. Epub 2016 Feb 8. PMID 26853526
- [Background] Hudnut-Beumler J, Po'e E, Barkin S. The Use of Social Media for Health Promotion in Hispanic Populations: A Scoping Systematic Review. JMIR Public Health Surveill. 2016 Jul 11;2(2):e32. doi: 10.2196/publichealth.5579. PMID 27400979
- [Background] JaKa MM, Haapala JL, Trapl ES, Kunin-Batson AS, Olson-Bullis BA, Heerman WJ, Berge JM, Moore SM, Matheson D, Sherwood NE. Reporting of treatment fidelity in behavioural paediatric obesity intervention trials: a systematic review. Obes Rev. 2016 Dec;17(12):1287-1300. doi: 10.1111/obr.12464. Epub 2016 Sep 9. PMID 27612933
- [Background] Heerman WJ, White RO, Hotop A, Omlung K, Armstrong S, Mathieu I, Sherwood NE, Barkin SL. A Tool Kit to Enhance the Informed Consent Process for Community-Engaged Pediatric Research. IRB. 2016 Sep-Oct;38(5):8-14. No abstract available. PMID 29442474
- [Background] Heerman WJ, Berge JM, Barkin SL. Mentoring of Early-Stage Investigators When Funding Is Tight: The Childhood Obesity Prevention and Treatment Research Experience. JAMA Pediatr. 2018 Jan 1;172(1):4-6. doi: 10.1001/jamapediatrics.2017.3396. No abstract available. PMID 29181507
- [Background] Heerman WJ, Lounds-Taylor J, Mitchell S, Barkin SL. Validity of the toddler feeding questionnaire for measuring parent authoritative and indulgent feeding practices which are associated with stress and health literacy among Latino parents of preschool children. Nutr Res. 2018 Jan;49:107-112. doi: 10.1016/j.nutres.2017.10.018. Epub 2017 Nov 3. PMID 29224793
- [Background] Heerman WJ, JaKa MM, Berge JM, Trapl ES, Sommer EC, Samuels LR, Jackson N, Haapala JL, Kunin-Batson AS, Olson-Bullis BA, Hardin HK, Sherwood NE, Barkin SL. The dose of behavioral interventions to prevent and treat childhood obesity: a systematic review and meta-regression. Int J Behav Nutr Phys Act. 2017 Nov 15;14(1):157. doi: 10.1186/s12966-017-0615-7. PMID 29141651
- [Background] Fletcher GE, Teeters L, Schlundt D, Bonnet K, Heerman WJ. Maternal conception of gestational weight gain among Latinas: A qualitative study. Health Psychol. 2018 Feb;37(2):132-138. doi: 10.1037/hea0000555. Epub 2017 Oct 2. PMID 28967775
- [Background] van Bakergem M, Sommer EC, Heerman WJ, Hipp JA, Barkin SL. Objective reports versus subjective perceptions of crime and their relationships to accelerometer-measured physical activity in Hispanic caretaker-child dyads. Prev Med. 2017 Feb;95 Suppl:S68-S74. doi: 10.1016/j.ypmed.2016.12.001. Epub 2016 Dec 6. PMID 27939263
- [Background] Barkin SL, Lamichhane AP, Banda JA, JaKa MM, Buchowski MS, Evenson KR, Bangdiwala SI, Pratt C, French SA, Stevens J. Parent's Physical Activity Associated With Preschooler Activity in Underserved Populations. Am J Prev Med. 2017 Apr;52(4):424-432. doi: 10.1016/j.amepre.2016.11.017. Epub 2017 Jan 9. PMID 28081998
- [Background] Heerman WJ, Taylor JL, Wallston KA, Barkin SL. Parenting Self-Efficacy, Parent Depression, and Healthy Childhood Behaviors in a Low-Income Minority Population: A Cross-Sectional Analysis. Matern Child Health J. 2017 May;21(5):1156-1165. doi: 10.1007/s10995-016-2214-7. PMID 28092060
- [Background] Oelsner KT, Guo Y, To SB, Non AL, Barkin SL. Maternal BMI as a predictor of methylation of obesity-related genes in saliva samples from preschool-age Hispanic children at-risk for obesity. BMC Genomics. 2017 Jan 9;18(1):57. doi: 10.1186/s12864-016-3473-9. PMID 28068899
- [Background] Stevens J, Pratt C, Boyington J, Nelson C, Truesdale KP, Ward DS, Lytle L, Sherwood NE, Robinson TN, Moore S, Barkin S, Cheung YK, Murray DM. Multilevel Interventions Targeting Obesity: Research Recommendations for Vulnerable Populations. Am J Prev Med. 2017 Jan;52(1):115-124. doi: 10.1016/j.amepre.2016.09.011. Epub 2016 Oct 26. PMID 28340973
- [Background] Heerman WJ, Mitchell SJ, Thompson J, Martin NC, Sommer EC, van Bakergem M, Taylor JL, Buchowski MS, Barkin SL. Parental perception of built environment characteristics and built environment use among Latino families: a cross-sectional study. BMC Public Health. 2016 Nov 22;16(1):1180. doi: 10.1186/s12889-016-3854-7. PMID 27876038
- [Background] Mathieu NP, Sommer EC, Mitchell SJ, Barkin SL. Urban Latino Families' Food Built Environment and Young Children's Produce Consumption. J Health Care Poor Underserved. 2016;27(4):1899-1908. doi: 10.1353/hpu.2016.0170. PMID 27818446
- [Background] Heerman WJ, White RO, Barkin SL. Advancing informed consent for vulnerable populations. Pediatrics. 2015 Mar;135(3):e562-4. doi: 10.1542/peds.2014-3041. No abstract available. PMID 25713286
- [Background] Ruiz RM, Sommer EC, Tracy D, Banda JA, Economos CD, JaKa MM, Evenson KR, Buchowski MS, Barkin SL. Novel patterns of physical activity in a large sample of preschool-aged children. BMC Public Health. 2018 Feb 13;18(1):242. doi: 10.1186/s12889-018-5135-0. PMID 29439704
- [Background] French SA, Sherwood NE, Mitchell NR, Fan Y. Park use is associated with less sedentary time among low-income parents and their preschool child: The NET-Works study. Prev Med Rep. 2016 Nov 10;5:7-12. doi: 10.1016/j.pmedr.2016.11.003. eCollection 2017 Mar. PMID 27872802
- [Background] Pratt CA, Boyington J, Esposito L, Pemberton VL, Bonds D, Kelley M, Yang S, Murray D, Stevens J. Childhood Obesity Prevention and Treatment Research (COPTR): interventions addressing multiple influences in childhood and adolescent obesity. Contemp Clin Trials. 2013 Nov;36(2):406-13. doi: 10.1016/j.cct.2013.08.010. Epub 2013 Aug 31. PMID 23999502
- [Background] Berge JM, Truesdale KP, Sherwood NE, Mitchell N, Heerman WJ, Barkin S, Matheson D, Levers-Landis CE, French SA. Beyond the dinner table: who's having breakfast, lunch and dinner family meals and which meals are associated with better diet quality and BMI in pre-school children? Public Health Nutr. 2017 Dec;20(18):3275-3284. doi: 10.1017/S1368980017002348. Epub 2017 Sep 14. PMID 28903804
- [Background] Cui Z, Truesdale KP, Robinson TN, Pemberton V, French SA, Escarfuller J, Casey TL, Hotop AM, Matheson D, Pratt CA, Lotas LJ, Po'e E, Andrisin S, Ward DS. Recruitment strategies for predominantly low-income, multi-racial/ethnic children and parents to 3-year community-based intervention trials: Childhood Obesity Prevention and Treatment Research (COPTR) Consortium. Trials. 2019 May 28;20(1):296. doi: 10.1186/s13063-019-3418-0. PMID 31138278
- [Background] Heerman WJ, Sommer EC, Slaughter JC, Samuels LR, Martin NC, Barkin SL. Predicting Early Emergence of Childhood Obesity in Underserved Preschoolers. J Pediatr. 2019 Oct;213:115-120. doi: 10.1016/j.jpeds.2019.06.031. Epub 2019 Jul 26. PMID 31353040
- [Background] Gesell SB, de la Haye K, Sommer EC, Saldana SJ, Barkin SL, Ip EH. Identifying Social Network Conditions that Facilitate Sedentary Behavior Change: The Benefit of Being a "Bridge" in a Group-based Intervention. Int J Environ Res Public Health. 2020 Jun 12;17(12):4197. doi: 10.3390/ijerph17124197. PMID 32545539
- [Background] Gesell SB, Sommer EC, Barkin SL. The 'GROW Social Network' datasets. Connections. 2020;40(1):123-128.
- [Background] LeCroy MN, Nicastro HL, Truesdale KP, Matheson DM, Ievers-Landis CE, Pratt CA, Jones S, Sherwood NE, Burgess LE, Robinson TN, Yang S, Stevens J. Dietary patterns and associations with BMI in low-income, ethnic minority youth in the USA according to baseline data from four randomised controlled trials. Br J Nutr. 2021 Jul 14;126(1):81-91. doi: 10.1017/S0007114520003852. Epub 2020 Sep 30. PMID 32993818
- [Background] Heerman WJ, Samuels LR, Barr L, Burgess LE, Hartmann KE, Barkin SL. The Effect of a General Healthy Lifestyle Intervention Delivered Around Pregnancy on Gestational Weight Gain and Infant Growth. Matern Child Health J. 2020 Nov;24(11):1404-1411. doi: 10.1007/s10995-020-02998-0. PMID 32815077
- [Background] Heerman WJ, Sommer EC, Qi A, Burgess LE, Mitchell SJ, Samuels LR, Martin NC, Barkin SL. Evaluating dose delivered of a behavioral intervention for childhood obesity prevention: a secondary analysis. BMC Public Health. 2020 Jun 8;20(1):885. doi: 10.1186/s12889-020-09020-w. PMID 32513226
- [Background] Heerman WJ, Wilkins CH, Barkin SL. Disseminating aggregate research findings to participants. Pediatr Res. 2021 Mar;89(4):714-715. doi: 10.1038/s41390-020-0995-2. Epub 2020 Jun 3. No abstract available. PMID 32492697
- [Background] Rushing A, Sommer EC, Zhao S, Po'e EK, Barkin SL. Salivary epigenetic biomarkers as predictors of emerging childhood obesity. BMC Med Genet. 2020 Feb 14;21(1):34. doi: 10.1186/s12881-020-0968-7. PMID 32059710
- [Background] Rachal SS, Heerman WJ, Sommer EC, Martin NC, Barkin SL. A longitudinal analysis of relationships between neighborhood context and underserved children's physical activity in a rapidly growing city. Prev Med Rep. 2021 Jun 11;23:101437. doi: 10.1016/j.pmedr.2021.101437. eCollection 2021 Sep. PMID 34178589
- [Background] Gesell SB, Barkin SL, Ip EH, Saldana SJ, Sommer EC, Valente TW, de la Haye K. Leveraging Emergent Social Networks to Reduce Sedentary Behavior in Low-Income Parents With Preschool-Aged Children. Sage Open. 2021 Jul-Sep;11(3):10.1177/21582440211031606. doi: 10.1177/21582440211031606. Epub 2021 Jul 23. PMID 37275840
- [Background] Tracy JD, Donnelly T, Sommer EC, Heerman WJ, Barkin SL, Buchowski MS. Identifying bedrest using waist-worn triaxial accelerometers in preschool children. PLoS One. 2021 Jan 28;16(1):e0246055. doi: 10.1371/journal.pone.0246055. eCollection 2021. PMID 33507967
- [Result] Barkin SL, Heerman WJ, Sommer EC, Martin NC, Buchowski MS, Schlundt D, Po'e EK, Burgess LE, Escarfuller J, Pratt C, Truesdale KP, Stevens J. Effect of a Behavioral Intervention for Underserved Preschool-Age Children on Change in Body Mass Index: A Randomized Clinical Trial. JAMA. 2018 Aug 7;320(5):450-460. doi: 10.1001/jama.2018.9128. PMID 30088008
- [Derived] Drengler A, Sommer EC, Sneed NM, McMahon E, Truesdale KP, Matheson D, Noerper TE, Samuels LR, Barkin SL, Heerman WJ. Federal Nutrition Assistance Programs and UltraProcessed Food Intake among Preschool-Aged Children. Curr Dev Nutr. 2025 Sep 27;9(11):107564. doi: 10.1016/j.cdnut.2025.107564. eCollection 2025 Nov. PMID 41189741
- [Derived] JaKa MM, Wood C, Veblen-Mortenson S, Moore SM, Matheson D, Stevens J, Atkins L, Michie S, Adegbite-Adeniyi C, Olayinka O, Po'e EK, Kelly AM, Nicastro H, Bangdiwala SI, Barkin SL, Pratt C, Robinson TN, Sherwood NE. Applying the Behavior Change Technique Taxonomy to Four Multicomponent Childhood Obesity Interventions. West J Nurs Res. 2021 May;43(5):468-477. doi: 10.1177/0193945920954782. Epub 2020 Sep 10. PMID 32909523